CLINICAL TRIAL: NCT02776371
Title: Modified Non-clarithromycin Triple Therapy in Eradicating Helicobacter Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016SDU-QILU-05
Record Dates: First submitted 2016-05-15; First posted 2016-05-18 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Helicobacter Pylori Eradication Rate
Keywords: Helicobacter pylori; Sequential therapy; Modified non-clarithromycin triple therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified non-clarithromycin triple therapy (Experimental): H.pylori infected patients treated with 10 mg rabeprazole twice a day, and 1g amoxicillin, 500 mg tinidazole three times a day for 14 days.
  Interventions: Drug: Modified non-clarithromycin triple therapy
- Sequential therapy (Active Comparator): H.pylori infected patients treated with 10 mg rabeprazole and 1 g amoxicillin, twice daily for 7 days, followed by 10 mg rabeprazole, 500 mg clarithromycin, and 500 mg tinidazole, twice daily for the next 7 days.
  Interventions: Drug: Sequential therapy

INTERVENTIONS:
Drug: Modified non-clarithromycin triple therapy — H. pylori infected patients treated with 10 mg rabeprazole twice a day, and 1g amoxicillin, 500 mg tinidazole three times a day for 14 days.
  Arms: Modified non-clarithromycin triple therapy
Drug: Sequential therapy — H. pylori infected patients treated with 10 mg rabeprazole and 1 g amoxicillin, twice daily for 7 days, followed by 10 mg rabeprazole, 500 mg clarithromycin, and 500 mg tinidazole, twice daily for the next 7 days.
  Arms: Sequential therapy

SUMMARY:
Helicobacter pylori (H. pylori) infects more than 50% of the population in the world(1), especially 47-66% in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were intend to undergo upper endoscopy for any purpose and volunteered to written inform consent.

Exclusion Criteria:

* negative in rapid urease test (RUT)
* previous standard eradication therapy for H. pylori;
* history of esophagectomy or gastrectomy;
* gastrointestinal malignancy;
* contraindications or allergic to study drugs;
* user of taking medicine that may affect the result of the study within 4 weeks (e.g., proton-pump inhibitors, H2-receptor antagonists, bismuth or antibiotics etc.);
* cardiopulmonary, hepatic or renal insufficiency, and/or severe current diseases or malignancy;
* pregnant or lactating women;
* participants of other trial within the past 3 months;
* unwilling or unable to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
the difference of eradication rates between 2 groups | 5 months

SECONDARY OUTCOMES:
the different rates of adverse events between 2 groups | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China